CLINICAL TRIAL: NCT02990897
Title: Pilot Study of Health Information Technology for Chronic Kidney Disease Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Lipika Samal, Associate Physician, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0
Record Dates: First submitted 2016-12-08; First posted 2016-12-13 (Estimated); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Chronic Kidney Disease
Keywords: Medical informatics; Quality of care; Referral
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (No Intervention): Patients with Stage 3,4, or 5 CKD who are randomized to the control arm will receive standard care.
- Intervention Group (Experimental): Patients with Stage 3,4, or 5 CKD who are randomized to the intervention group will receive care from a physician who has been exposed to the intervention: a clinical decision support message. This clinical decision support message shows the patient's risk of kidney failure over the next 5 years.
  Interventions: Behavioral: clinical decision support message

INTERVENTIONS:
Behavioral: clinical decision support message — The intervention patient's physician is shown an estimate of the patient's 5 year risk of ESRD with a link for further information.
  Arms: Intervention Group

SUMMARY:
Researchers now know that treating chronic kidney disease (CKD) in its early stages can prevent dialysis and reduce heart problems that go along with kidney disease. Computerized tools may help primary care doctors to diagnose the disease earlier and computer reminders may help doctors to prescribe the best treatments. In this project the investigators will test computer reminders in primary care clinics to see if they improve treatment of early chronic kidney disease and to see if it can promote referral to nephrology.

DETAILED DESCRIPTION:
The investigators are conducting a randomized trial to determine the effect of a health information technology (HIT) application to calculate risk progression of end stage renal disease (ESRD). The primary outcome is the completion of the necessary tests for the risk prediction model (urine albumin to creatinine ratio, serum calcium, serum phosphate, serum albumin, and serum bicarbonate) for CKD patients in primary care. Secondary outcomes will include nephrology referrals, doubling of serum creatinine, initiation of hemodialysis, and primary care provider (PCP) satisfaction. In the analysis, all patients over the age of 18 who have a visit with one of physicians involved in the trial during the intervention period will be eligible and patients with stage 3-5 CKD will be included. Physicians are the subjects in this study, as the intervention is a behavioral intervention for physicians. The physicians' patients will not actively be recruited and will only indirectly be affected by the study. The application creates blocks of patient appointments for each physician and randomly assigns patients to intervention and control arms within these blocks.

ELIGIBILITY:
Inclusion Criteria:

* patients who are 18 years or older
* patients of primary care providers who are included in the study
* patients with CKD (defined as two estimated glomerular filtration rate (GFR) values under 60 mL/min per 1.73 m^2 90 days apart)

Exclusion Criteria:

* patients without CKD (defined as two GFR values under 60 mL/min per 1.73 m^2 90 days apart)
* patients under the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2015-12; Primary Completion 2017-01 (Actual); Study Completion 2022-07-14 (Actual)

PRIMARY OUTCOMES:
Laboratory tests completed | 6 months following primary care visit
  Dichotomous measure of whether laboratory tests necessary to calculate the risk prediction model (urine albumin to creatinine ratio, serum calcium, serum phosphate, serum albumin, and serum bicarbonate) were resulted in the electronic health record for patients who did not previously have all of these tests done in the prior year.

SECONDARY OUTCOMES:
Urine microalbumin to creatinine ratio test completed | 6 months following primary care visit
  Dichotomous measure of whether urine microalbumin to creatinine ratio test was completed for patients who did not previously have these tests done in the prior year.
Referral of patient from PCP to nephrologist | 6 months following primary care visit
  Dichotomous measure of whether a patient was seen by a nephrologist for patients who did not previously have these tests done in the prior year.

CONTACTS AND LOCATIONS:
Overall Officials: Lipika Samal, MD, MPH, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- North Shore Physicians Group, Danvers, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Samal L, D'Amore JD, Gannon MP, Kilgallon JL, Charles JP, Mann DM, Siegel LC, Burdge K, Shaykevich S, Lipsitz S, Waikar SS, Bates DW, Wright A. Impact of Kidney Failure Risk Prediction Clinical Decision Support on Monitoring and Referral in Primary Care Management of CKD: A Randomized Pragmatic Clinical Trial. Kidney Med. 2022 May 28;4(7):100493. doi: 10.1016/j.xkme.2022.100493. eCollection 2022 Jul. PMID 35866010